CLINICAL TRIAL: NCT03627234
Title: Same Day Discharge vs. Overnight Stay After Minimally Invasive Hysterectomy: A Randomized Controlled Trial
Brief Title: Same Day Discharge vs. Overnight Stay After Hysterectomy
Acronym: SDD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the institution
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041832
Record Dates: First submitted 2018-07-30; First posted 2018-08-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Satisfaction; Safety Issues; Quality of Life
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Same Day Discharge (Experimental): Same day discharge after hysterectomy is the standard of care at George Washington University Hospital.
  Interventions: Behavioral: Same Day Discharge
- Overnight stay (Experimental): Overnight stay is not the standard of care at George Washington University Hospital. It is being used as an experimental condition.
  Interventions: Behavioral: Overnight Stay

INTERVENTIONS:
Behavioral: Same Day Discharge — Patients will be randomized to same day discharge
  Arms: Same Day Discharge
Behavioral: Overnight Stay — Patients will be randomized to stay overnight
  Arms: Overnight stay

SUMMARY:
In this study patients are randomized between same-day discharge and overnight stay after undergoing a minimally invasive hysterectomy or myomectomy. The goal is to both compare patients' satisfaction and safety and quality of life (QOL) as well as financial consequences between the two groups.

The investigators hope to demonstrate that same-day discharge is safe and feasible for most patients with the same level of satisfaction and safety and QOL compared to overnight stay. And also the investigators seek to determine which demographic, medical, social and intra-operative factors influence duration of admission, satisfaction, safety and QOL.

DETAILED DESCRIPTION:
1. Subject recruitment and consent: Subject recruitment will take place in the GW MFA outpatient clinic for the MIGS surgeons among patients desiring a myomectomy or a hysterectomy for a benign gynecologic reason (heavy bleeding, fibroids, pelvic pain) without comorbidities that require overnight stay (as decided by their provider). Interested subjects will be counseled and consented by a member of the research team. If the subjects choose to participate the consent form will be signed at that time or if the subjects need more time to consider participation the consent form will be signed at the pre-operative visit.
2. At the pre-operative visit, computer-generated randomization will be used to assign patients to

   A) Discharge the day of surgery (before midnight on the day of surgery) OR B) Discharge after an overnight stay.

   Patients will be informed about their assigned group during this visit to be able to prepare their discharge and recovery period with care-takers at home. Participants will complete the health-related quality of life (HrQoL) questionnaire EQ-5D before surgery as a baseline measurement and complete a survey including basic demographic information (detailed prior).
3. Study participants will then undergo a minimally invasive hysterectomy or myomectomy by one of the highly experienced minimally invasive gynecologists using a standard technique. Their approaches to hysterectomy and myomectomy are similar and according to the normal standard of care.
4. In case of protocol deviation by participants,the investigators will record why the participants decided to deviate from the protocol to be able to identify factors that influence length of hospital stay. The investigators will conduct an intention-to-treat analysis to correct for these protocol deviations. The investigators will counsel patients thoroughly to try to minimize the number of protocol deviations.
5. Hospital (operative and pathology reports) and clinical (clinical visit notes) reports will be reviewed to compare baseline demographics, preoperative hemoglobin, past surgical history, past medical history, comorbidities, operative time, case end time, estimated blood loss, uterine weight and complications between the same-day discharge and overnight stay group.
6. Patients will complete the HrQoL questionnaire on days 0, 1, 2, 4 and 7 using the self- completed EQ-5D.
7. Hospital and ED notes will be checked for unexpected postoperative visits, re-evaluations and re-admissions.
8. At their postoperative visit 2 weeks after their surgery patients will be asked to complete the surgical satisfaction questionnaire (SSQ-8) and to score feelings of safety regarding the timing of their discharge on a scale from 0-10

ELIGIBILITY:
Inclusion Criteria:

* Myomectomy or hysterectomy planned for a benign gynecologic reason. (This means that there is no evidence of, or concern for, malignancy in the cervix, uterus, tubes or ovaries. Benign gynecologic reasons to have a hysterectomy include fibroids, abnormal uterine bleeding, endometriosis, and pelvic pain.)
* Patient is scheduled to have surgery with one of the minimally invasive gynecologic surgeons at GWUH. (Dr. Moawad, Dr. Marfori, Dr. Abi Khalil or Dr. Vargas)
* Patient is planned for a robotic assisted total laparoscopic hysterectomy (RA-TLH), a total laparoscopic hysterectomy (TLH), a robotic assisted laparoscopic myomectomy (RA-myomectomy) or a laparoscopic myomectomy.
* Patient is capable of informed consent.
* Patient is capable of completing the questionnaires.
* Patient must be between 18 and 65 years of age.

Exclusion Criteria:

* Myomectomy or hysterectomy is indicated for malignancy.
* Procedure is anything other than RA-TLH, TLH, RA-myomectomy or a laparoscopic myomectomy.
* Surgeon is not one of the minimally invasive surgeons at GWUH.
* Surgery is scheduled for a hospital other than GWUH.
* Patient is less than 18 years of age or greater than 65.
* Patient is not capable of informed consent.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender females
Enrollment: 0 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction as measured by the Surgical Satisfaction Scale | 2 weeks
  Patient satisfaction with Same day discharge vs overnight stay. This will be measured using the Surgical Satisfaction Questionnaire The SSQ is an 8-item questionnaire, with responses recorded on a 5-point Likert type scale with responses from 0 "Very Unsatisfied" to 4 "Very Satisfied." The mean average of the 8 scores is being multiplied by 25 (the questionnaire is considered incomplete if more than 2 items are not answered), yielding a potential range of scores from 0 to 100. The higher the score is, the greater the degree of surgical satisfaction. Items 1 and 2 are used to calculate the Pain subscale; items 3, 4, and 5 are used for the Return to baseline subscale: and items 6, 7, and 8 are used for the Global satisfaction subscale. The questionnaire will be administered after surgery (day 10-14 postoperatively) at their postoperative visit at the clinic.

SECONDARY OUTCOMES:
Health Related Quality of life | 6 weeks
  The quality of life that patients report using the Health related quality of life EuroQuol group, the Netherlands. The EQ-5D has 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The instrument has been shown to be valid and reliable for use in a wide range of health conditions and can be administered daily

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States